CLINICAL TRIAL: NCT00042861
Title: A Phase I Pharmacologic Trial Of Infusional UCN-01 Given With A Weekly Schedule Of 5-Fluorouracil And Leucovorin
Brief Title: UCN-01, Fluorouracil, and Leucovorin in Treating Patients With Metastatic or Unresectable Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069478; NCI-NAVY-01-04; NCI-5535; NCI-02-C-0222; NCT00039637 (obsolete NCT alias)
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2003-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — 7-hydroxystaurosporine; Fluorouracil; Leucovorin

INTERVENTIONS:
Drug: 7-hydroxystaurosporine
Drug: fluorouracil
Drug: leucovorin calcium

SUMMARY:
RATIONALE: UCN-01 may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining UCN-01 with chemotherapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining UCN-01, fluorouracil, and leucovorin in treating patients who have metastatic or unresectable solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of fluorouracil when given in combination with UCN-01 and leucovorin calcium in patients with metastatic or unresectable solid tumors.
* Determine the clinical toxic effects of this regimen in these patients.
* Determine the pharmacokinetics of these drugs in these patients.
* Correlate, if possible, the pharmacokinetics of these drugs with clinical toxicity in these patients.
* Assess the pharmacodynamic effects of these drugs in these patients.
* Assess any clinical activity of this regimen in patients with measurable disease.

OUTLINE: This is a dose-escalation study of fluorouracil (5-FU).

Patients receive leucovorin calcium (CF) IV over 2 hours and 5-FU IV (at the midpoint of CF administration) on day 1, followed by UCN-01 IV over 36-72 hours, on weeks 1-3. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of 5-FU until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. The recommended phase II dose (RPIID) is defined as the dose preceding the MTD. At least 6 additional patients are treated at the RPIID.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study within 16 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor that is metastatic or unresectable and for which no standard curative or palliative measures exist or are effective
* No brain metastases or primary CNS malignancy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* AST and ALT no greater than 3 times upper limit of normal

Renal

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No known active coronary artery disease

Pulmonary

* No pulmonary dysfunction

Other

* HIV negative
* No history of unusually severe and/or prolonged toxicity during prior therapy with fluorouracil (5-FU) or 5-FU prodrugs
* No diabetes mellitus requiring insulin or oral hypoglycemic therapy
* No ongoing or active infection requiring IV antibiotics
* No other serious concurrent medical illness that would preclude study
* No psychiatric illness or social situations that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 4 weeks since prior immunotherapy and recovered
* No concurrent cytokines during the first course of therapy

Chemotherapy

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy

* No concurrent systemic corticosteroids

Radiotherapy

* At least 2 weeks since prior radiotherapy and recovered
* No prior pulmonary or mediastinal radiation exceeding 40 Gy

Surgery

* Recovered from prior surgery

Other

* No other concurrent investigational agents
* No concurrent cimetidine
* No concurrent sorivudine or brivudine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-08

CONTACTS AND LOCATIONS:
Overall Officials: Jean L. Grem, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States